CLINICAL TRIAL: NCT03950323
Title: Intra-parotid Facial Nerve by MRI Tractography: Clinical vs Radiologic Description in Parotid Tumors
Brief Title: Intra-parotid Facial Nerve Tractography
Acronym: R-PO19053
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO19053
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Parotid Tumor
Keywords: Parotidetomy; Tractography; Facial nerve; Facial palsy; Tumor of parotid gland
MeSH Terms: conditions — Parotid Neoplasms; Facial Paralysis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients operated on for parotid tumor (Experimental): All consecutive patients operated on for parotid tumor.
  Interventions: Radiation: MRI with Facial nerve tractography

INTERVENTIONS:
Radiation: MRI with Facial nerve tractography — MRI with Facial nerve tractography in addition to T1 imaging, T1 gadolinium imaging and T2 imaging.

SUMMARY:
The aim of the study is to evaluate concordance between the facial nerve's path in the parotid evaluated by radiologist in preoperatively and the facial nerve's path in the parotid evaluated by surgeon in peroperatively.

DETAILED DESCRIPTION:
Surgery is the main treatment for parotid tumol, benign or malignant pathologies. The procedure requires a trunk search and a facial nerve dissection along its intraparotid length. This intervention entails a risk of facial paralysis.

MRI tractography is a new imaging technique that can characterize nerve fibers and their path.

The interest would be to allow the surgeon to best prepare the parotidectomy by locating the tumor in relation to the trunk and all the branches of the facial nerve.

ELIGIBILITY:
inclusion criteria :

* Major patient
* Patient with initial parotid mass or recurrent
* Parotidian mass with surgical indication
* Benign or malignant
* With or without preoperative facial paralysis
* Patients consenting the protocol

exclusion criteria :

* Parotidian masses without surgical indication
* Patient with a classic contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-12-24 (Estimated); Study Completion 2021-06-24 (Estimated)

PRIMARY OUTCOMES:
Facial nerve's path | Day 0
  Relations between the facial nerve's (the facial nerve's trunk s and the facial nerve's dissections) and the parotid gland will be studied. The nerve will be
  * in front of the mass or behind the mass
  * below the mass or above the mass
  * outside the mass or inside the mass

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France